CLINICAL TRIAL: NCT01506401
Title: The Oscillation for ARDS Treated Early (OSCILLATE) Trial
Brief Title: The Oscillation for Acute Respiratory Distress Syndrome (ARDS) Treated Early (OSCILLATE) Trial
Acronym: OSCILLATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolment halted by Steering Committee on advice from Data Monitoring Committee.
Sponsor: Canadian Critical Care Trials Group (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT94829; ISRCTN87124254 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2011-12-14; First posted 2012-01-10 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2012-09

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: ARDS; ventilator-induced lung injury; lung protective ventilation; high frequency oscillation
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Ventilation (Active Comparator): Low tidal volumes, relatively high PEEP.
  Interventions: Procedure: Lung Protective Ventilation
- High Frequency Oscillation (Experimental): Open-lung strategy for high frequency oscillation.
  Interventions: Device: SensorMedics 3100B High Frequency Oscillatory Ventilator

INTERVENTIONS:
Device: SensorMedics 3100B High Frequency Oscillatory Ventilator — High Frequency Oscillation
  Arms: High Frequency Oscillation
Procedure: Lung Protective Ventilation — Tidal Volume 6ml/kg; plateau pressure < or = 35cmH20; Prescribed PEEP/FiO2 chart
  Arms: Conventional Ventilation

SUMMARY:
What is the effect of early high frequency oscillation (HFO) versus a lung-protective conventional ventilation (CV) strategy (using HFO only as rescue therapy), on all-cause hospital mortality among patients with severe early acute respiratory distress syndrome (ARDS)?

DETAILED DESCRIPTION:
High frequency oscillation is theoretically ideal for lung protection. Based on a strong physiological rationale, rapidly expanding use internationally, and promising results in early small RCTS, a definitive RCT to establish the impact of HFO versus current conventional ventilation on mortality is needed. We have completed a pilot multicentre RCT in preparation for this trial, with goals of investigating patient recruitment, protocol acceptance, and crossover rates. The pilot study met all objectives including recruitment that exceeded expectations (94 patients), and very good adherence to protocol. Results of the multinational OSCILLATE Trial will establish the impact of HFO versus conventional ventilation on mortality rates among adults with severe ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of respiratory failure, with fewer than 2 weeks of new pulmonary symptoms;
* Endotracheal intubation or tracheostomy;
* Hypoxaemia - defined as a partial pressure of oxygen in arterial blood (PaO2)/fraction of inspired oxygen (FiO2) less than or equal to 200mmHg on FiO2 greater than or equal to 0.5, regardless of positive end expiratory pressure (PEEP)
* Bilateral alveolar consolidation (airspace disease) seen on frontal chest radiograph

In addition, to qualify for randomization, patients are assessed on the following ventilator settings:

* Mode: pressure control or volume control or pressure support
* FiO2 greater than 0.6 (or higher if necessary to keep pulse oximetric saturation [SpO2] greater than 90%)
* PEEP greater than 10 cm H2O (or greater if necessary to keep SpO2 greater than 90%)
* Tidal volume 6 ml/kg predicted body weight (PBW)

After at least 30 minutes on these settings, we sample arterial blood to assess oxygenation. If PaO2 is less than or equal to 200 mmHg, the patient qualifies for randomization; if PaO2/FiO2 greater than 200 mmHg, standardized hypoxaemia assessments are repeated at least once daily for the following 72 hours (providing eligibility criteria are still met).

Exclusion Criteria:

* Remaining duration of mechanical ventilation less than 48 hours, as judged by the attending physician
* Primary cause of acute respiratory failure judged by attending physician to be circulatory overload due to, for example, congestive heart failure, hyper-resuscitation, or need for dialysis
* Suspected pulmonary haemorrhage syndrome
* Lack of commitment to ongoing life support (note that this does not include the presence of a "Do Not Resuscitate" order alone, if there is a commitment to ongoing life support
* Aged less than 16 years or greater than 85 years
* Weight less than 35 kg
* Severe chronic respiratory disease, as indicated by any of:
* Baseline forced expiratory volume in one second (FEV1) less than 20 ml/kg predicted body weight
* Pre-existing chronic interstitial lung disease with chronic interstitial infiltration on chest x-ray
* Documented chronic carbon dioxide (CO2) retention (partial pressure of carbon dioxide in arterial blood [PaCO2] less than 50 mmHg) and/or chronic hypoxaemia(PaO2 less than 55 mmHg on FiO2=0.21)
* Chronic restrictive, obstructive, neuromuscular, chest wall or pulmonary vascular disease resulting in severe exercise restriction (e.g., unable to climb stairs or perform household duties), secondary polycythaemia, severe pulmonary hypertension (mean pulmonary arterial pressure [PAP] greater than 40 mmHg), or ventilator dependency
* Morbid obesity - defined as greater than 1 kg/cm body height
* Underlying pre-existing condition with expected 6-month mortality greater than 50%
* Neurological conditions with risk of intracranial hypertension (where hypercapnia should be avoided)
* Neuromuscular disease that will result in prolonged need for mechanical ventilation, including (but not limited to):
* Guillain Barre syndrome
* Cervical spinal cord injury
* Previous randomization in this trial
* All inclusion criteria present for greater than 73 hours in study intensive care unit (ICU)
* On HFO at the time of screening

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
All-cause hospital mortality | Randomised patients will be ventilated according to their assigned ventilation strategy for up to 60 days, until they die on the ventilator or are successfully (for >24 hours) liberated from mechanical ventilation.
  all-cause hospital mortality

SECONDARY OUTCOMES:
Mortality at other time-points | Duration of hospitalization (ICU discharge, 60 days)
  mortality at other time-points (ICU discharge, 60 days)
Barotrauma | ICU discharge or 60 days
  Barotrauma
Organ Dysfunction | Duration of hospitalization or 60 days
  Organ Dysfunction
Duration of mechanical ventilation | Duration of hospitalization or 60 days
  Duration of mechanical ventilation
Duration of ICU & Hospital Stay | Duration of hospitalization which may exceed 60 days
  Duration of ICU & Hospital Stay
Quality of Life at 6 months | 6 months post randomization
  Quality of Life at 6 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Niall D Ferguson, MD, MSc, Principal Investigator — University of Toronto; Maureen O Meade, MD, MSc, Principal Investigator — McMaster University
Locations (38):
- United States (8):
  - Denver Health Medical Centre, Denver, Colorado
  - Orlando Regional Medical Centre, Orlando, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Hospital of the University ofPennsylvania, Philadelphia, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas HSC, Houston, Texas
  - Texas A&M HSC College of Medicine, Scott & White Hospital, Temple, Texas
- Canada (24):
  - Peter Lougheed Centre/Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Medical Centre, Edmonton, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver Island Health Research Centre, Victoria, British Columbia
  - Health Sciences Centre, Winnipeg, Winnipeg, Manitoba
  - Royal Victoria Hospital, Barrie, Ontario
  - St. Joseph's Healthcare, McMaster University, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - University of Western Ontario - University Hospital, London, Ontario
  - University of Western Ontario - Victoria Hospital, London, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St Josephs, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - William Osler Health Centre, Toronto, Ontario
  - Maisonneuve Rosemont, Montreal, Quebec
  - Centre Hosptialier de liUniersite de Montreal - CHUM- Saint Luc, Montreal, Quebec
  - Patrick Bellemare, Montreal, Quebec
  - Hopital de l'Enfant-Jesus, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
- Chile (2):
  - Clinica Las Lilas, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
- Deenanath Mangeshkar Hospital & Research Centre, Pune, India
- Saudi Arabia (3):
  - King Faisal Specialist Hospital & Research Centre, Jeddah
  - King Fahad National Guard Hospital, Riyadh
  - Riyadh Armed Forces, Riyadh

REFERENCES:
- [Derived] Arabi YM, Cook DJ, Zhou Q, Smith O, Hand L, Turgeon AF, Matte A, Mehta S, Graham R, Brierley K, Adhikari NK, Meade MO, Ferguson ND; Canadian Critical Care Trials Group. Characteristics and Outcomes of Eligible Nonenrolled Patients in a Mechanical Ventilation Trial of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1306-13. doi: 10.1164/rccm.201501-0172OC. PMID 26192398
- [Derived] Ferguson ND, Cook DJ, Guyatt GH, Mehta S, Hand L, Austin P, Zhou Q, Matte A, Walter SD, Lamontagne F, Granton JT, Arabi YM, Arroliga AC, Stewart TE, Slutsky AS, Meade MO; OSCILLATE Trial Investigators; Canadian Critical Care Trials Group. High-frequency oscillation in early acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):795-805. doi: 10.1056/NEJMoa1215554. Epub 2013 Jan 22. PMID 23339639